CLINICAL TRIAL: NCT07095101
Title: Effect and Cost-effectiveness of Smartphone-based Behavioural Intervention on Orofacial Pain
Brief Title: ePROPP - eHealth for Preventing and Reducing Orofacial Pain in the Population
Acronym: ePROPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: Folktandvården Skåne AB (Other)
Responsible Party: Principal Investigator, Birgitta Haggman Henriksson, Professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dnr 2024-05598-01
Record Dates: First submitted 2025-07-14; First posted 2025-07-31 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Joint Disorder; Temporomandibular Disorders (TMDs)
Keywords: Temporomandibular Disorders (TMDs); Myalgia; Facial Pain; Behavior therapy; Telemedicine; Digital health; Occlusal splints; Cost-effectiveness analysis; Bruxism; Mobile applications; Cognitive Behavioral Therapy
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia; Facial Pain; Bruxism | interventions — Occlusal Splints

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mobistudy Application (Experimental): Treatment with mobile application
  Interventions: Behavioral: Mobistudy Application
- Occlusal splint (Active Comparator): Treatment with an occlusal splint
  Interventions: Device: Occlusal splint
- Waiting list (No Intervention): Waiting list followed by delayed intervention with mobile application

INTERVENTIONS:
Behavioral: Mobistudy Application — Treatment with mobile application
  Arms: Mobistudy Application
Device: Occlusal splint — Treatment with an occlusal splint
  Arms: Occlusal splint

SUMMARY:
Pain in the orofacial region has a 10% prevalence in the general population and health care providers are therefore expected to encounter these patients on a daily basis. Chronic orofacial pain often presents as jaw pain related to overload of the jaw muscles and temporomandibular joints. The aim of this study is to evaluate the effectiveness of a smartphone-based behavioural intervention (Ecological Momentary Intervention, EMI) grounded in Cognitive Behavioural Therapy (CBT), compared to standard treatment with an occlusal splint and a waiting list control group.

DETAILED DESCRIPTION:
The World Health Organization (WHO) emphasizes oral health as a key indicator of overall wellbeing. Poor oral health, especially when associated with pain, severely impacts individuals by reducing their quality of life. Orofacial pain is the third most common chronic pain, after knee and neck/back pain, and affects more than 10% of the adult population worldwide. In common with other chronic pain conditions, orofacial pain is a multi-factorial condition involving biological, psychological, and social factors - all encompassed in the biopsychosocial model. Contributing factors to pain, such as stress and anxiety are increasing, highlighting the need to identify and manage patients to counteract this growing problem. One potential risk factor for orofacial pain is muscle and joint overload due to stress-related tooth clenching and grinding. It is therefore important to evaluate and modify behaviours related to such overload.

Shortage of resources results in many patients not receiving treatment. In addition to the suffering experienced by affected individuals, chronic pain also significantly impacts family members, and leads to increased healthcare costs and a substantial societal burden.

Effective treatments, such as cognitive behavioural therapy (CBT), are available, but time-consuming, requiring repeated visits to care providers. Consequently, the incorporation of eHealth solutions utilizing mobile technology and internet-based therapy has been recommended. The implementation of eHealth, defined as "the use of information and communications technology in support of health and health-related fields" is advocated by the WHO to "accelerate global attainment of health and wellbeing". The recent development of smartphone and internet-based applications offers a promising avenue for cost-effectiveness and equity in health care

Traditional treatment of orofacial pain with oral splints requires repeated dental visits and incur significant costs together with additional technician costs for splint fabrication. A digital behavioural intervention could offer a drastically more cost-effective solution, reduce patients' suffering and the number of treatment visits, thereby easing the burden on the current waiting lists for patients with orofacial pain that in many regions can be a year or more. The project will investigate whether digital behavioural intervention can serve as a cost-effective alternative to traditional occlusal splint therapy for managing orofacial pain. By integrating real-time data collection and intervention, patients can be offered personalized, accessible treatment that seamlessly integrate into daily life. The availability of cost-effective eHealth solutions is especially relevant in regions with limited access to health care due to geographical distances or shortage of health care providers. Moreover, eHealth medical care can also be invaluable in situations for patients who are homebound for any reason.

This project aims to gain unique knowledge into the core mechanisms of pain and evaluate a novel multimodal person-centred eHealth approach for management of orofacial pain.

The overarching goal is to develop and evaluate a cost-effective eHealth tool for management of orofacial pain in collaboration with health care providers, facilitating large scale implementation in the population. The non-inferiority hypothesis: Treatment with a smartphone based behavioural intervention is not inferior to treatment with occlusal splint.

The superiority hypothesis: Compared to waiting list, a smartphone based behavioural intervention can reduce orofacial pain.

The results from this project can enable a broad implementation of an eHealth treatment that conserves resources, helping to address the current resource shortages in healthcare.

ELIGIBILITY:
Inclusion criteria

* Chronic orofacial pain, duration ≥3 months with a diagnosis of Myalgia according to the brief DC/TMD.
* Patients will be included even if they have one or more additional DC/TMD diagnoses
* Regular smartphone users
* Understanding written and spoken Swedish
* Age ≥ 18 years

Exclusion criteria

* Other orofacial non-TMD pain conditions
* Cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-22 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | From enrolment to 3 month follow-up
  Pain level will be assessed using the Numeric rating Scale (NRS, a scale ranging from 0 (no pain) to 10 (worst pain imaginable). A 30% reduction in pain according to the NRS is considered a significant effect.

SECONDARY OUTCOMES:
Cost-effectiveness | From enrolment to 3 month follow-up
  Cost-effectiveness will be assessed using direct and indirect costs to calculate total societal costs for the two different interventions
Stress-levels | From enrolment to 3 month follow-up
  Assessment of stress will be done using the Perceived stress-scale (PSS-10) which yields a total score from 0 to 40, calculated by summing responses to 10 items, each scored on a 5-point Likert scale (0 = never to 4 = very often).
Changes in general well-being | From enrolment to 3 month follow-up
  Assessment of general wellbeing will be done with Patient Health Questionnaire (PHQ-4) which combines two 2-item scales: the PHQ-2 (depression) and the GAD-2 (anxiety). Each question is scored on a 4-point Likert scale (0-3), and the total score is the sum of all four items Higher scores indicate a greater severity of symptoms.
Correlation between pain and overload | From enrolment to 3 month follow-up
  During the first 3 days of using the mobistudy application, the relation between muscluskeletal overload and TMD-pain will be assessed..
  Assessment of overload with Ecological momentary assessment of self-reported overload will be correlated (Spearman's correlated) to pain intensity using the Numeric rating Scale (NRS), a scale ranging from 0 (no pain) to 10 (worst pain imaginable).

OTHER OUTCOMES:
Coping | From enrolment to 3 month follow-up
  Coping will be assessed with the Brief Resilience Coping Scale (BRCS-4) using a 5-point Likert scale for each item, ranging from "Does not describe me at all" to "Describes me very well". The total score is calculated by summing the responses to all four items. Higher scores indicate a greater tendency toward resilient coping.
Headache | From enrolment to 3 month follow-up
  Assessment with the Headache screening questionnaire (HSQ). The HSQ aims to identify individuals who might have migraine or tension type headache by assessing headache characteristics across four domains: frequency, duration, characteristics, and symptoms.
Widespread pain | From enrolment to 3 month follow-up
  Widespread pain will be assessed by a pain manikin.

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta Häggman-Henrikson, DDS, PhD, Principal Investigator — Malmö University

IPD SHARING:
Plan to Share IPD: No
Restrictions related to sensitive personal data and ethical approval

REFERENCES:
- [Background] Stanisic N, Do CT, Skarping S, Chrcanovic B, Bracci A, Manfredini D, Haggman-Henrikson B. Smartphone application to report awake bruxism: Development and testing of the Swedish version and a pilot study to evaluate family history in young adults and their parents. J Oral Rehabil. 2024 Jan;51(1):188-195. doi: 10.1111/joor.13515. Epub 2023 May 29. PMID 37210658
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331
- [Background] Haggman-Henrikson B, Liv P, Ilgunas A, Visscher CM, Lobbezoo F, Durham J, Lovgren A. Increasing gender differences in the prevalence and chronification of orofacial pain in the population. Pain. 2020 Aug;161(8):1768-1775. doi: 10.1097/j.pain.0000000000001872. Epub 2020 Mar 16. PMID 32701837
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934